CLINICAL TRIAL: NCT03124381
Title: A Multi-Center, Evaluator Blinded, Randomized Clinical Study to Evaluate the Efficacy and Tolerance of Two Acne Treatment Regimens on Subjects With Mild to Moderate Acne Vulgaris
Brief Title: A Study to Evaluate the Efficacy and Tolerance of 2 Acne Treatment Regimens on Subjects With Mild to Moderate Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PS-170103145529-SACT
Record Dates: First submitted 2017-04-03; First posted 2017-04-21 (Actual); Results first posted 2018-11-09 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluator-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Acne Mask (Active Comparator): Cleanser, Acne Mask
  Interventions: Device: Cleanser, Acne Mask
- Gel-Cream + Acne Mask (Experimental): Cleanser, Gel-Cream, Acne Mask
  Interventions: Device: Cleanser, Gel-Cream, Acne Mask

INTERVENTIONS:
Device: Cleanser, Acne Mask — A facial cleanser will be used twice daily (morning and evening). The light therapy mask will be used for 10 minutes in the evening after washing/drying the face.
  Other Names: Light Therapy Mask
  Arms: Acne Mask
Device: Cleanser, Gel-Cream, Acne Mask — A facial cleanser will be used twice daily (morning and evening). In the evening after cleansing, the gel-cream will be applied full face and allowed to dry before the light therapy mask is used for 10 minutes.
  Other Names: Light Therapy Mask; Light Therapy Topical Gel-Cream
  Arms: Gel-Cream + Acne Mask

SUMMARY:
This study will compare two different acne treatment regimens for the treatment of acne. Half of participants will receive a cleanser and a light therapy mask, while half of the participants will receive a cleanser, a light therapy topical gel-cream, and a light therapy mask.

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic skin disease involving blockage and/or inflammation of the hair follicles and their accompany sebaceous glands.

Research has shown the benefits of red and blue light therapy in the treatment of mild to moderate acne, with red and blue light shown to target acne-causing bacteria and have an effect on inflammation reduction.

Light-based therapies have been used successfully to treat dermatological conditions since the early 1900s, with various parts of the electromagnetic spectrum (i.e. ultraviolet [UV], visible, near-infrared, etc.) demonstrating different benefits. Light-emitting diodes (LEDs) offer delivery of light to the skin in a gentler manner as compared to light delivered by lasers, primarily due to the lower energy output. It has been reported that LEDs do not deliver enough power to damage tissues and do not have the same risk of accidental eye damage that lasers do. Visible-LED light therapy has been deemed a non-significant risk by the U.S. Food and Drug Administration (FDA) and has been approved for use in humans.

It is well established in the literature that visible light penetration into the epidermal and dermal layers of human skin is primarily governed by absorption and scattering events, with the latter being the more impactful of the two. Visible light penetration into human skin can be increased by reducing scattering. This can be accomplished by temporary hydrogen bonding disruption, which leads to the reversible rearrangement of epidermal and dermal structures that cause scattering. Glycerol (i.e. glycerin) is hypothesized to generate the level of hydrogen bonding disruption described above, and therefore will be investigated in the present study.

This study will look to evaluate and then compare the acne clearing efficacy and tolerance of two different acne treatment regimens - a cleanser used with a currently marketed red and blue light acne light therapy mask alone vs. the cleanser used with the same mask in conjunction with a light therapy topical gel-cream - to determine the efficacy of these treatments and then to assess if the efficacy of the light therapy mask used with the topical gel-cream treatment is non-inferior to the mask alone in the reduction of lesions in mild to moderate acne. If non-inferiority is demonstrated, the mask with topical gel-cream treatment will be further assessed for its superiority to the mask alone.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate facial acne
* Has 10-100 blackheads/whiteheads, 10-50 pimples, no cysts, and up to 2 large, hard, painful bumps (nodules)
* Able to read, write, speak, and understand English
* In general good health
* Must agree to practice a medically acceptable form of birth control.
* Intends to complete the study and willing to follow all study instructions.

Exclusion Criteria:

* Very sensitive skin or allergies/sensitivity to skincare products or the test product ingredients.
* Has a light or photosensitivity disorder or another medical condition that could increase risk to the subject or confuse the study results
* Is using medication that makes skin more sensitive to light
* Has severe acne or a pre-existing facial skin condition other than mild to moderate acne
* has an immune deficiency disorder
* has been using a product or medication that the stuff investigator determines will increase health risk to the subject or confuse the study results
* Females that are pregnant, nursing, or planning to become pregnant
* Males with a female partner who is pregnant or planning to become pregnant
* Has excessive facial hair
* Is participating in another study within past 4 weeks
* Is related to the Sponsor, Investigator, or Study Site

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2017-04-08 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Bucko, D.O., Principal Investigator — Academic Dermatology Associates; Lily Jiang, Ph.D., Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (2):
- United States (2):
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Thomas J. Stephens and Associates, Inc., Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashkenazi H, Malik Z, Harth Y, Nitzan Y. Eradication of Propionibacterium acnes by its endogenic porphyrins after illumination with high intensity blue light. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):17-24. doi: 10.1111/j.1574-695X.2003.tb00644.x. PMID 12589953
- [Background] Kjeldstad B. Photoinactivation of Propionibacterium acnes by near-ultraviolet light. Z Naturforsch C Biosci. 1984 Mar-Apr;39(3-4):300-2. doi: 10.1515/znc-1984-3-417. PMID 6730638
- [Background] Roelandts R. A new light on Niels Finsen, a century after his Nobel Prize. Photodermatol Photoimmunol Photomed. 2005 Jun;21(3):115-7. doi: 10.1111/j.1600-0781.2005.00160.x. No abstract available. PMID 15888126
- [Background] Barolet D. Light-emitting diodes (LEDs) in dermatology. Semin Cutan Med Surg. 2008 Dec;27(4):227-38. doi: 10.1016/j.sder.2008.08.003. PMID 19150294
- [Background] Salomatina E, Jiang B, Novak J, Yaroslavsky AN. Optical properties of normal and cancerous human skin in the visible and near-infrared spectral range. J Biomed Opt. 2006 Nov-Dec;11(6):064026. doi: 10.1117/1.2398928. PMID 17212549
- [Background] Bashkatov, AN, et al. Optical properties of melanin in the skin and skin-like phantoms. Proc. of SPIE, 4162: 219-226, 2000.
- [Background] Bashkatov, AN, et al. Optical properties of human skin, subcutaneous and mucous tissues in the wavelength range from 400 to 2000 nm. J Phys D: Appl Phys, 38: 2543-2555, 2005.
- [Background] Jacques SL. Optical properties of biological tissues: a review. Phys Med Biol. 2013 Jun 7;58(11):R37-61. doi: 10.1088/0031-9155/58/11/R37. Epub 2013 May 10. PMID 23666068
- [Background] Lamouche G, Kennedy BF, Kennedy KM, Bisaillon CE, Curatolo A, Campbell G, Pazos V, Sampson DD. Review of tissue simulating phantoms with controllable optical, mechanical and structural properties for use in optical coherence tomography. Biomed Opt Express. 2012 Jun 1;3(6):1381-98. doi: 10.1364/BOE.3.001381. Epub 2012 May 15. PMID 22741083
- [Background] Pogue BW, Patterson MS. Review of tissue simulating phantoms for optical spectroscopy, imaging and dosimetry. J Biomed Opt. 2006 Jul-Aug;11(4):041102. doi: 10.1117/1.2335429. PMID 16965130
- [Background] Hirshburg J, Choi B, Nelson JS, Yeh AT. Correlation between collagen solubility and skin optical clearing using sugars. Lasers Surg Med. 2007 Feb;39(2):140-4. doi: 10.1002/lsm.20417. PMID 17311267
- [Background] Wiegand, B, Luedtke, K, Rapp, SR. Acne Profile. Johnson & Johnson, One Johnson & Johnson Plaza, New Brunswick, NJ 08933-7003, assignee. Patent US 2006/0008484 A1. 12 Jan. 2006. Print.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Started | 65 | 61
Completed | 56 | 55
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Non-Compliance with Study Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gel-Cream + Acne Mask | Acne Mask | Total
Number analyzed (Participants) | 65 | 61 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.8 (6.03) | 20.0 (7.65) | 19.4 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 70
  Male | 27 | 29 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 23 | 48
  Not Hispanic or Latino | 40 | 38 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 47 | 47 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Skin Sensitivity [Count of Participants; unit: Participants] — Self-perceived skin sensitivity. Do you consider your skin to be sensitive...none of the time, some of the time, most of the time, all of the time
  Participants
    None of the Time | 38 | 40 | 78
    Some of the Time | 21 | 18 | 39
    Most of the Time | 6 | 1 | 7
    All of the Time | 0 | 2 | 2
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Description:Measure of skin type characteristics, including sensitivity to burning/tanning. Ranging from I to VI, where I = White; very fair; red or blonde hair; blue eyes; freckles; Always burns easily; never tans and VI = Black; black hair, black eyes, black skin; Never burns; deeply pigmented
  Participants
    I | 0 | 0 | 0
    II | 24 | 28 | 52
    III | 18 | 14 | 32
    IV | 12 | 10 | 22
    V | 10 | 6 | 16
    VI | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Global Face Total Lesion Count - Percent Change - Baseline to Week 12
Description: Percent change from baseline in global face total lesion count at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population was used, including all subjects with data for this time point. Missing values were imputed by carrying forward the last observed post-baseline score. There was no post-baseline data to carry forward for three subjects.
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Percent Change in Lesions | -42.64 (31.817) | -47.80 (30.209)
Statistical Analysis 1: Comparison: Gel-Cream + Acne Mask vs Acne Mask; Non-inferiority test performed after significance vs. baseline confirmed for each cell. The null hypothesis for the non-inferiority test was H0: A-B≥15%, where A and B are the mean percent change at Week 12 of global face total acne lesion count of the Gel-Cream + Acne Mask cell and Acne Mask cell, respectively; Test type: Non-Inferiority — Non-inferiority concluded if the upper bound of the two-sided 95% confidence interval (based on ANCOVA) is less than 15 percentage points. Terms for treatment, gender, center as factors and baseline as covariate; Mean Difference (Net) = 3.19, 95% CI 2-sided [-7.04 to 13.42], Standard Error of Mean 5.164
Statistical Analysis 2: Comparison: Gel-Cream + Acne Mask vs Acne Mask; Superiority test performed after non-inferiority confirmed as described above. The null hypothesis for the superiority test was H0: A-B = 0, where A and B are the mean percent change at Week 12 of global face total acne lesion count of the Acne Mask and the Gel-Cream + Acne Mask cell, respectively; Test type: Superiority — Superiority concluded if the upper bound of the two-sided 95% confidence interval of the treatment difference is less than 0. Terms for treatment, gender, and center as factors and baseline score as covariate; p = 0.538, ANCOVA; Mean Difference (Net) = 3.19, 95% CI 2-sided [-7.04 to 13.42], Standard Error of Mean 5.164

2. Secondary Outcome: Global Face Total Lesion Count - Percent Change - Baseline to Week 2
Description: Percent change from baseline in global face total lesion count at Week 2
Time Frame: Baseline and Week 2
Population: Intent-to-treat population was used, including all subjects with data for this time point. The number may be less than the total due to subject withdrawal prior to this time point or missed visits/evaluations.
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Percent Change in Lesions | -24.16 (25.646) | -27.97 (21.330)

3. Secondary Outcome: Global Face Total Lesion Count - Percent Change - Baseline to Week 4
Description: Percent change from baseline in global face total lesion count at Week 4
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Percent Change in Lesions | -29.78 (27.388) | -38.25 (22.729)

4. Secondary Outcome: Global Face Total Lesion Count - Percent Change - Baseline to Week 8
Description: Percent change from baseline in global face total lesion count at Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Percent Change in Lesions | -39.81 (26.192) | -45.86 (23.369)

5. Secondary Outcome: Global Face Total Lesion Count - Percent Change From Baseline to the Mean of All Visits
Description: Global face total lesion counts are averaged across all applicable post-baseline visits (Week 2, Week 4, Week 8, and Week 12). Percent change from baseline to the mean is then calculated.
Time Frame: Baseline to Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Percent Change in Lesions | -33.68 (24.212) | -39.79 (20.754)

6. Secondary Outcome: Global Face Total Lesion Count - Percent Change From Baseline to the Mean of Week 2 and Week 4
Description: Global face total lesion counts are averaged across Week 2 and Week 4. Percent change from baseline to the mean is then calculated.
Time Frame: Baseline to Week 2 and Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Percent Change in Lesions | -26.95 (24.419) | -33.01 (19.648)

7. Secondary Outcome: Global Face Total Lesion Count - Percent Change From Baseline to the Mean of Week 4 and Week 8
Description: Global face total lesion counts are averaged across Week 4 and Week 8. Percent change from baseline to the mean is then calculated.
Time Frame: Baseline to Week 4 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Percent Change in Lesions | -34.34 (25.438) | -42.09 (21.082)

8. Secondary Outcome: Global Face Total Lesion Count - Percent Change From Baseline to the Mean of Week 8 and Week 12
Description: Global face total lesion counts are averaged across Week 8 and Week 12. Percent change from baseline to the mean is then calculated.
Time Frame: Baseline to Week 8 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change in Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 58 | 55
Percent Change in Lesions | -41.73 (27.472) | -47.25 (46.201)

9. Secondary Outcome: Global Face Open Comedones Count - Week 2
Description: Open comedones count on global face - Week 2
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Open Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Open Comedones | 8.1 (10.68) | 5.6 (6.41)

10. Secondary Outcome: Global Face Open Comedones Count - Week 4
Description: Open comedones count on global face - Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Open Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Open Comedones | 7.9 (10.37) | 5.3 (6.27)

11. Secondary Outcome: Global Face Open Comedones Count - Week 8
Description: Open comedones count on global face - Week 8
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Open Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Open Comedones | 5.1 (7.83) | 4.5 (6.03)

12. Secondary Outcome: Global Face Open Comedones Count - Week 12
Description: Open comedones count on global face - Week 12
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Open Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Open Comedones | 3.6 (5.2) | 3.7 (6.31)

13. Secondary Outcome: Global Face Closed Comedones Count - Week 2
Description: Closed comedones count on global face - Week 2
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Closed Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Closed Comedones | 14.7 (10.66) | 12.7 (9.41)

14. Secondary Outcome: Global Face Closed Comedones Count - Week 4
Description: Closed comedones count on global face - Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Closed Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Closed Comedones | 14.1 (11.69) | 10.9 (7.01)

15. Secondary Outcome: Global Face Closed Comedones Count - Week 8
Description: Closed comedones count on global face - Week 8
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Closed Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Closed Comedones | 12.7 (10.38) | 10.3 (7.05)

16. Secondary Outcome: Global Face Closed Comedones Count - Week 12
Description: Closed comedones count on global face - Week 12
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Closed Comedones
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Closed Comedones | 11.9 (10.01) | 10.2 (9.00)

17. Secondary Outcome: Global Face Inflammatory Lesion Count - Week 2
Description: Papules and pustules counted together
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Inflammatory Lesions | 12.1 (8.23) | 10.3 (5.24)

18. Secondary Outcome: Global Face Inflammatory Lesion Count - Week 4
Description: Papules and pustules counted together
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Inflammatory Lesions | 10.8 (7.56) | 9.1 (6.15)

19. Secondary Outcome: Global Face Inflammatory Lesion Count - Week 8
Description: Papules and pustules counted together
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Inflammatory Lesions | 9.9 (6.85) | 7.8 (5.07)

20. Secondary Outcome: Global Face Inflammatory Lesion Count - Week 12
Description: Papules and pustules counted together
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Inflammatory Lesions | 9.7 (7.19) | 7.7 (6.44)

21. Secondary Outcome: Global Face Non-Inflammatory Lesion Count - Week 2
Description: Sum of open comedones and closed comedones
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Non-inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Non-inflammatory Lesions | 22.7 (15.94) | 18.3 (11.74)

22. Secondary Outcome: Global Face Non-Inflammatory Lesion Count - Week 4
Description: Sum of open comedones and closed comedones
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Non-inflammatory lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Non-inflammatory lesions | 22.0 (16.39) | 16.2 (10.51)

23. Secondary Outcome: Global Face Non-Inflammatory Lesion Count - Week 8
Description: Sum of open comedones and closed comedones
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Non-inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Non-inflammatory Lesions | 17.8 (13.92) | 14.8 (10.68)

24. Secondary Outcome: Global Face Non-Inflammatory Lesion Count - Week 12
Description: Sum of open comedones and closed comedones
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Non-inflammatory Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Non-inflammatory Lesions | 15.6 (12.92) | 14.0 (13.39)

25. Secondary Outcome: Global Face Total Lesion Count - Week 2
Description: Sum of inflammatory and non-inflammatory lesions
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Lesions | 34.8 (19.30) | 28.6 (13.10)

26. Secondary Outcome: Global Face Total Lesion Count - Week 4
Description: Sum of inflammatory and non-inflammatory lesions
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Lesions | 32.8 (20.10) | 25.2 (13.53)

27. Secondary Outcome: Global Face Total Lesion Count - Week 8
Description: Sum of inflammatory and non-inflammatory lesions
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Lesions | 27.7 (17.41) | 22.5 (13.95)

28. Secondary Outcome: Global Face Total Lesion Count - Week 12
Description: Sum of inflammatory and non-inflammatory lesions
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Lesions | 25.3 (17.56) | 21.7 (17.58)

29. Secondary Outcome: Investigator Global Acne Assessment - Week 1
Description: Investigator Global Acne Assessment using Modified Cooke's Scale - Week 1. Modified Cooke's scale ranges from 0 = clear/no acne to 5 = very severe acne. Half-points are allowed.
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 64 | 60
Units on a scale | 2.29 (0.444) | 2.27 (0.427)

30. Secondary Outcome: Investigator Global Acne Assessment - Week 2
Description: Investigator Global Acne Assessment using Modified Cooke's Scale - Week 2. Modified Cooke's scale ranges from 0 = clear/no acne to 5 = very severe acne. Half-points are allowed.
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Units on a scale | 2.17 (0.500) | 2.06 (0.470)

31. Secondary Outcome: Investigator Global Acne Assessment - Week 4
Description: Investigator Global Acne Assessment using Modified Cooke's Scale - Week 4. Modified Cooke's scale ranges from 0 = clear/no acne to 5 = very severe acne. Half-points are allowed.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Units on a scale | 2.00 (0.587) | 1.90 (0.583)

32. Secondary Outcome: Investigator Global Acne Assessment - Week 8
Description: Investigator Global Acne Assessment using Modified Cooke's Scale - Week 8. Modified Cooke's scale ranges from 0 = clear/no acne to 5 = very severe acne. Half-points are allowed.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Units on a scale | 1.84 (0.669) | 1.73 (0.600)

33. Secondary Outcome: Investigator Global Acne Assessment - Week 12
Description: Investigator Global Acne Assessment using Modified Cooke's Scale - Week 12. Modified Cooke's scale ranges from 0 = clear/no acne to 5 = very severe acne. Half-points are allowed.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Units on a scale | 1.64 (0.724) | 1.64 (0.589)

34. Secondary Outcome: Overall Redness of Inflammatory Lesions - Week 1
Description: Additional investigator efficacy assessment. 0-9 scale where 0 = no redness associated with the inflammatory lesions; 9 = overall, inflammatory lesions exhibit severe degree of redness
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 64 | 60
Units on a scale | 4.88 (1.222) | 5.05 (1.278)

35. Secondary Outcome: Overall Redness of Inflammatory Lesions - Week 2
Description: as for outcome 34
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Units on a scale | 4.65 (1.183) | 4.74 (1.202)

36. Secondary Outcome: Overall Redness of Inflammatory Lesions - Week 4
Description: as for outcome 34
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Units on a scale | 4.49 (1.291) | 4.41 (1.318)

37. Secondary Outcome: Overall Redness of Inflammatory Lesions - Week 8
Description: as for outcome 34
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Units on a scale | 4.30 (1.278) | 4.25 (1.446)

38. Secondary Outcome: Overall Redness of Inflammatory Lesions - Week 12
Description: as for outcome 34
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Units on a scale | 3.96 (1.346) | 3.97 (1.282)

39. Secondary Outcome: Overall Size of Inflammatory Lesions - Week 1
Description: Additional investigator efficacy assessment. 0-9 scale where 0 = no longer visible; 9 = overall size is very large
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 64 | 60
Units on a scale | 4.58 (1.298) | 4.83 (1.371)

40. Secondary Outcome: Overall Size of Inflammatory Lesions - Week 2
Description: Additional investigator efficacy assessment. Additional investigator efficacy assessment. 0-9 scale where 0 = no longer visible; 9 = overall size is very large
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 63 | 60
Units on a scale | 4.17 (1.129) | 4.56 (1.222)

41. Secondary Outcome: Overall Size of Inflammatory Lesions - Week 4
Description: as for outcome 40
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 62 | 56
Units on a scale | 4.07 (1.273) | 4.15 (1.408)

42. Secondary Outcome: Overall Size of Inflammatory Lesions - Week 8
Description: as for outcome 40
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 57 | 55
Units on a scale | 3.88 (1.290) | 3.85 (1.606)

43. Secondary Outcome: Overall Size of Inflammatory Lesions - Week 12
Description: as for outcome 40
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
Number analyzed (Participants) | 56 | 55
Units on a scale | 3.67 (1.305) | 3.59 (1.411)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent through subject's last study procedure (Week 12 unless terminated early). Serious adverse events (SAE) reported to the site were also reportable within 30 days of last procedure/visit and longer if considered study-related; there was no specific cut-off date for this reporting, but AEs/SAEs are shown in this posting for a collection period of 1 year from last subject's visit (the time of this posting).
Description: The Investigator or a designee interviewed subjects for changes in health/medication at each visit, documenting any reported adverse events.
Arm/Group | Gel-Cream + Acne Mask | Acne Mask
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/61
Other Adverse Events (participants affected / at risk) | 0/65 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide Sponsor 60 days to review any publication (unless expedited review requested); if includes Sponsor's confidential info, written Sponsor approval is required. Sponsor may require another 60 days' delay to file patent app. If multicenter, PI agrees 1st publication is joint publication. If joint publication not submitted within 24 months of study end or Sponsor confirms there will be no joint publication, PI may publish the results individually following previous guidelines.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT03124381/SAP_000.pdf
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03124381/Prot_001.pdf